## PROSPECTIVE STUDY INVESTIGATING THE OPTIMAL DURATION OF INDWELLING URINARY CATHETER FOLLOWING INFRAPERITONEAL COLORECTAL SURGERY AND ROLE OF POSTOPERATIVE ALPHA-BLOCKADE

**Protocol:** Version 3, 11/30/2012

**Lead Investigator:** Phillip Fleshner, MD

Phillip Fleshner, MD Division of Colorectal Surgery Cedars-Sinai Medical Center

## **PROTOCOL**

| Protocol No./ Title: | Prospective study investigating the optimal duration of indwelling urinary catheter following infraperitoneal colorectal surgery and role of postoperative alpha-blockade | |
|---|---|---|
| Study Rationale | The purpose of this study is to evaluate whether a postoperative pelvic colorectal patient can safely have an indwelling catheter removed on postoperative day one with the addition of a study medication, without a statistically significant difference in the incidence of urinary retention compared to the standard, accepted approach of delayed removal. | |
| Study Population: | Determine the incidence of retention of two groups. A control group of 72 hours catheterization (Group 1) to 24 hours catheterization plus medication (Group 2) to potentially reduce retention. | |
| | <ul> <li>Data Description: Non-inferiority study p<sub>A</sub>=0.15, p<sub>B</sub>=0.15, d=0.15 (tolerance).</li> <li>We would like to test 1) If Group 2 is non-inferior to Group 1 (2 is not worse than 1).</li> </ul> | |
| | Power Analysis and Sample Size Calculation: | |
| | A sample size for 80% power is 71 per group. This would be a total of 142. | |
| | Two group test of equivalence in proportions | |
| | Test significance level, a (one-sided) Standard proportion, ps Equivalence limit difference, | 0.050<br>0.150 |
| | p <sub>T</sub> - p <sub>S</sub> , D <sub>0</sub> Test expected proportion, p <sub>T</sub> Expected difference, p <sub>T</sub> - p <sub>S</sub> , D <sub>1</sub> Power (%) n per group | 0.150<br>0.150<br>0.000<br>80<br>71 |
| Hypothesis | Early removal of a urinary catheter in postoperative infraperitoneal colorectal surgery patients will experience a similar incidence of acute urinary retention than delayed removal, will likely have a lower incidence of clinically important urinary tract infections, and experience improvement in quality of life measures. | |
| Study Design: | Single-center, randomized, prospective study. Pacatheter removal group will be given 1 mg prazo pharmacy will be responsible for the distribution when indicated. The study drug will be given 6 l removal in Group 2 patients. | sin orally (per os). The of the medication |

| Primary Efficacy<br>Endpoint: | Acute urinary retention (Re-catheterization) |
|---|---|
| Secondary | 1. Urinary tract infection (>10 <sup>5</sup> CFU/mL with symptoms) |
| <b>Endpoints:</b> | 2. Cardiopulmonary complications |
| | 3. Surgical site infections |
| | 4. Anastomotic leaks |
| | 5. Quality of life |
| | 6. Length of postoperative stay |
| | 7. Volume of retained urine if re-catheterized (Bladder Scan) |
| | 8. Adverse side effects from treatment drug |
| Safety Endpoints: | Receiving care patient would have otherwise received. |
| Sample size: | With a sample size of 71 patients per group for a total of 142 patients, this study will have 80% power to detect a statistically significant difference between acute urinary retention in patients with urinary catheter removal 24 hours postoperatively compared to 72 hours postoperatively. |
| Interim Analysis | There will be an interim analysis after 71 patients enrolled (half the study group) |
| Key Inclusion<br>Criteria: | 1. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form; |
| | 2. Males or females, >18 years of age inclusive at the time of study screening; |
| | 3. American Society of Anesthesiologists (ASA) Class I-III; |
| | 4. Infraperitoneal colorectal surgery (open and/or laparoscopic); |
| | 5. Elective Surgery |
| Key Exclusion<br>Criteria | 1. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures; |
| | 2. Children <18; |
| | 3. No perioperative antibiotics; |
| | 4. Past or current urinary tract malignancy; |
| | 5. Urinary catheter inserted before surgery; |
| | 6. Chronic kidney insufficiency with Creatinine> 2 |
| | 7. Diagnosis of benign prostatic hyperplasia |

| | 8. Chronic urinary infections |
|---|---|
| | • |
| | 9. Neurogenic bladder |
| | 10. History of enter vesicle fistula |
| | 11. Pregnancy |
| | 12. Prior surgery of the lower urinary tract |
| | 13. Epidural |
| | 14. Perioperative ureteral stents |
| | After randomization: |
| | 1. Catheter pulled out inadvertently; |
| | 2. Postoperative complications requiring prolonged monitoring of urine output |
| | 3. Postoperative complications requiring early reoperation |
| Treatment | Patients will be assigned into one of three groups: |
| Regimen/ Duration: | |
| | Group 2 – randomized to receive prazosin <b>6 hours prior to catheter removal</b> and removal of urinary catheter 24 hours postoperatively |
| Treatment Failure/<br>Discontinuation<br>Criteria: | Patients will be discontinued from the trial at any time as a result of any other event that in the opinion of the investigator warrants discontinuation from the trial. |
| | Additionally, patients will be excluded after randomization if: |
| | 1. Catheter pulled out inadvertently; |
| | 2. Postoperative complications requiring prolonged monitoring of urine output; |
| | 3. Postoperative complications requiring early reoperation |

## 2. SCHEDULE OF EVENTS

| | <del>-</del> |
|-----------------------------------------|--------------|
| | Group 1: |
| | Delayed |
| | Catheter |
| | removal |
| Visit Number | Admission |
| Informed Consent | |
| Demographics | |
| Height | |
| Medical History <sup>1</sup> | |
| Inclusion/ Exclusion Criteria | |
| Review | |
| Previous /Concomitant | |
| Medications | |
| Physical Exam <sup>2</sup> | |
| Vital Signs <sup>3</sup> | |
| Body Weight | |
| Adverse Events <sup>4</sup> | |
| Quality of Life Assessment <sup>5</sup> | ✓ |
| Hospital Discharge or Early | ./ |
| Termination Visit <sup>6</sup> | · |

- 1. Medical History obtained at index admission including: Hypertension, Lung Disease, Diabetes
- 2. Comprehensive physical exam performed at index admission
- 3. Vital Signs (systolic and diastolic blood pressure, heart rate, respiration rate, and temperature) at index admission.
- 4. Adverse events (AEs) will be recorded at every visit post screening. AEs will be followed until resolution.
- 5. Quality of Life assessment will be performed on last hospital day prior to discharge (Appendix A)
- 6. Early Termination visits are used when a patient withdraws from the study (i.e., prior to hospital discharge).

| | Group 2: Prazosin and early catheter removal |
|---|---|
| Visit Number | Admission |
| Informed Consent | |
| Demographics | |
| Height | |
| Medical History <sup>1</sup> | |
| Inclusion/ Exclusion Criteria<br>Review | |
| Previous /Concomitant<br>Medications | |
| Physical Exam <sup>2</sup> | |
| Vital Signs <sup>3</sup> | |
| Body Weight | |
| Adverse Events <sup>4</sup> | |
| Quality of Life Assessment <sup>5</sup> | ✓ |
| Hospital Discharge or Early<br>Termination Visit <sup>6</sup> | ✓ |

- 1. Medical History obtained at index admission including: Hypertension, Lung Disease, Diabetes
- 2. Comprehensive physical exam performed at index admission
- 3. Vital Signs (systolic and diastolic blood pressure, heart rate, respiration rate, and temperature) at index admission.
- 4. Adverse events (AEs) will be recorded at every visit post screening. AEs will be followed until resolution.
- 5. Quality of Life assessment will be performed on last hospital day prior to discharge (Appendix A)
- 6. Early Termination visits are used when a patient withdraws from the study (i.e., prior to hospital discharge).

| Postoperative Data Open or Laparoscopic Reason for surgery (benign or cancer) Type of Surgery (LAR, APR, IPAA, etc) ASA Score TMN stage Metastatic Lymph Nodes Total Mesorectal Excision Level of anastomosis (<5 cm from anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative Blood Loss (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> Quality of Life <sup>2</sup> | |
|---|---|
| Open or Laparoscopic Reason for surgery (benign or cancer) Type of Surgery (LAR, APR, IPAA, etc) ASA Score TMN stage Metastatic Lymph Nodes Total Mesorectal Excision Level of anastomosis (<5 cm from anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative Blood Loss (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | |
| Reason for surgery (benign or cancer) Type of Surgery (LAR, APR, IPAA, etc) ASA Score TMN stage Metastatic Lymph Nodes Total Mesorectal Excision Level of anastomosis (<5 cm from anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative Blood Loss (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | Postoperative Data |
| Type of Surgery (LAR, APR, IPAA, etc) ASA Score TMN stage Metastatic Lymph Nodes Total Mesorectal Excision Level of anastomosis (<5 cm from anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | Open or Laparoscopic |
| IPAA, etc) ASA Score TMN stage Metastatic Lymph Nodes Total Mesorectal Excision Level of anastomosis (<5 cm from anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | = |
| TMN stage Metastatic Lymph Nodes Total Mesorectal Excision Level of anastomosis (<5 cm from anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | |
| Metastatic Lymph Nodes Total Mesorectal Excision Level of anastomosis (<5 cm from anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | ASA Score |
| Total Mesorectal Excision Level of anastomosis (<5 cm from anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | TMN stage |
| Level of anastomosis (<5 cm from anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | Metastatic Lymph Nodes |
| anal verge) Neoadjuvant chemotherapy Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative Blood Loss (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | Total Mesorectal Excision |
| Neoadjuvant radiation therapy Intraoperative Fluid Volume (mL) Intraoperative Blood Loss (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | * |
| Intraoperative Fluid Volume (mL) Intraoperative Blood Loss (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | Neoadjuvant chemotherapy |
| Intraoperative Blood Loss (mL) Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | Neoadjuvant radiation therapy |
| Intraoperative/Postoperative Blood Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | Intraoperative Fluid Volume (mL) |
| Transfusion Bowel preparation Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | Intraoperative Blood Loss (mL) |
| Diverting stoma Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | 1 1 |
| Antibiotic therapy >24 hours postoperatively Morphine equivalent (mg) <sup>1</sup> | Bowel preparation |
| postoperatively Morphine equivalent (mg) <sup>1</sup> | Diverting stoma |
| · · · | ± • |
| Quality of Life <sup>2</sup> | Morphine equivalent (mg) <sup>1</sup> |
| | Quality of Life <sup>2</sup> |

- Morphine equivalent: 7 mg ≈ 1 mg hydromorphone
   Quality of Life: obtained on last day of hospitalization

| | Group 1 | Group 2 |
|----------------------------------------------------------|---------|---------|
| Endpoints | | |
| Acute urinary retention <sup>1</sup> (recatheterization) | | |
| Bladder scan volume (mL) | | |
| Symptomatic urinary tract infection <sup>2</sup> | | |
| Cardiopulmonary complications | | |
| Surgical site infection | | |
| Anastomotic Leak | | |
| Adverse side effects | | |
| Overall complication rate | | |
| Post-void residual (mL) | | |

- 1. Acute urinary retention defined as the inability to void despite urge and attempt, and/or the inability to void within 8 hours post-removal of the catheter.
- 2. Dysuria and >10<sup>5</sup> CFU/mL on urine culture